CLINICAL TRIAL: NCT03582371
Title: Effect of an Aqua Stand-Up Paddle Program on Postural Instability in Parkinson's Disease
Brief Title: Aqua Stand-Up Paddle Balance Effect in Parkinson's Disease (AquaSUP PARK)
Acronym: AquaSUP PARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FLABEAU Olivier (Other)
Responsible Party: Sponsor-Investigator, FLABEAU Olivier, Hospital practitionner, Centre Hospitalier de la côte Basque
Organization: Centre Hospitalier de la côte Basque (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P-2018/01
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease; Rehabilitation
Keywords: Parkinson's Disease; Rehabilitation; Balance; Aquatic therapy; Stand Up Paddle
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Proof of concept. Study of non-inferiority, prospective, monocentric, randomized, controlled (Aqua SUP vs physiotherapy), in blind treatment compared to applied treatment.
Who Masked: Outcomes Assessor
Masking Description: Patients will be scored Mini-Balance evaluation System Test by blinded investigators, before and after AquaSup or Physiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqua SUP (Experimental): Patients in the Aqua SUP group will benefit from a 1 hour Aqua SUP session, twice a week, for 8 weeks in a therapeutic pool.
  Interventions: Procedure: Stand-Up Paddle Rehabilitation
- Physiotherapy (Active Comparator): Patients in the control group will receive a conventional physiotherapy session of 1 hour, twice a week, for 8 weeks.
  Interventions: Procedure: Physiotherapy Rehabilitation

INTERVENTIONS:
Procedure: Stand-Up Paddle Rehabilitation — Patients in the Aqua SUP group will benefit from a 1 hour Aqua SUP session, twice a week, for 8 weeks in a therapeutic pool.
  Arms: Aqua SUP
Procedure: Physiotherapy Rehabilitation — Patients in the control group will receive a conventional physiotherapy session of 1 hour, twice a week, for 8 weeks.
  Arms: Physiotherapy

SUMMARY:
Postural instability is associated with falls and a decreased quality of life in Parkinson's disease (PD). Evidence supports physical activity rather than levodopa for postural instability management. Considering the proven effects of the Stand-up Paddle (SUP) activity on postural instability in sedentary people, the investigators wanted to develop this aquatic activity in a swimming pool on static conditions (Aqua SUP) for PD patients. The objective is to assess the postural instability change by measuring the Mini-Balance Evaluation Systems Test (miniBESTest) after 8 weeks of Aqua SUP compared to physiotherapy in PD patients with baseline postural instability.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a relentless neurodegenerative disorder leading to functional impairment with postural instability. Postural instability is associated with an increased risk of falling and a decreased quality of life, and levodopa therapy may only have little effect on balance. Evidence supports physiotherapy and physical activity as an alternative treatment for postural instability in PD. Several types of physical activity have been tested in PD which target different specificities of rehabilitation such as stretching, muscle strengthening, balance, occupational therapy, cueing, treadmill training, with contrasting data regarding postural instability. The investigators want to develop an innovative physical activity with specific focus on the management of the postural instability in PD patients. Stand-up Paddle (SUP) is an aquatic sport improving postural instability in sedentary people that may be practiced in a swimming pool with static conditions for safety (Aqua SUP).

In order to assess the effect on postural instability, PD patients with baseline postural instability will be scored by Mini-Balance Evaluation Systems Test (miniBESTest) before and after 8 weeks of Aqua SUP practice and compared to physiotherapy according to a randomized controlled trial with non-inferiority design.

Patients will be clinically assessed at baseline regarding the primary outcome miniBESTest and secondary outcome measures. A secondary visit will take place at 2 months after inclusion (Aqua SUP versus physiotherapy). A tertiary visit will be completed at 6 months after inclusion to assess long term effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 to 80 years of age.
* Patients suffering from idiopathic Parkinson's Disease according to the criteria of the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic.
* Presence of balance disorder : Stage Hoehn and Yahr 2.5 to 4.
* Motor level stable, without change of treatment in last 6 weeks
* Subjects affiliated to a social security scheme or beneficiary of an equivalent scheme
* Subjects are volunteers with their signed consent

Exclusion Criteria:

* Patients suffering from disabling neurological conditions other than IPD. Patients with progressive psychiatric pathologies.
* Patients with significant cognitive impairment (MMS <24).
* Presence of orthopedic problems incompatible with the practice of Aqua SUP.
* Medical advice against the practice of endurance exercise and muscle building.
* Patients with history or presence of cardiovascular or respiratory conditions, or patients who answered "yes" to any of the items in the Revised Physical Activity Readiness Questionnaire (Q-AAP).
* Patients with a condition which is deemed incompatible with the therapeutic pool: uncontrolled vesico-sphincteric disorder, aquaphobia, deterioration of the skin condition (wound, eschar, ulcer).
* Persons subject to decision making support (eg. legal guardianship or conservator).
* Patients in the process of participating in another study.
* Pregnant woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Mini-Balance Evaluation System Score variation | Change from baseline Mini-Balance Evaluation Systems Test at 2 months.
  Mini-Balance Evaluation System Test : Postural instability with falling risk evaluation, 14 items quoted 0 (severe) to 2 (normal). Total score recorded : minimum =0 Maximum =28. Higher values represent a better outcome

SECONDARY OUTCOMES:
Movement Disorder Society - Unified Parkinson's Disease rating Scale III score variation | Change from baseline Movement Disorder Society - Unified Parkinson's Disease rating Scale III at 2 months
  Movement Disorder Society - Unified Parkinson's Disease rating Scale III : Motor symptoms evaluation, 18 items quoted 0 (normal) to 4 (severe). Total score recorded : minimum =0 Maximum =72. Higher values represent a worse outcome
Berg Balance Scale score variation | Change from baseline Berg Balance Scale at 2 months
  Berg Balance Scale test : Balance and posture evaluation, 14 items quoted 0(normal) to 3 (severe). Total score recorded : Minimum=0 Maximum = 42. Higher values represent a worse outcome
Mini-Mental State Examination score variation | Change from baseline Mini-Mental State Examination: at 2 months
  Mini-Mental State Examination test : Cognitice capacity evaluation, 6 items evaluated. Total score recorded : Minimum = 0 Maximum = 30 . Higher values represent a better outcome
Modified Timed Up and Go score variation | Change from baseline Modified Modified Timed Up and Go at 2 months
  Modified Timed Up and Go Test : Functionnal capacity evaluation, Timing Walking test. Higher values represent a worse outcome
Global Mobility Task score variation | Change from baseline Global Mobility Task at 2 months
  Global Mobility Task Test : Functionnal capacity evaluation; 5 items quoted 0(normal) to 4 (severe). Total score recorded : Minimum=0 Maximum = 20. Higher values represent a worse outcome
2 minutes walking test score variation | Change from baseline 2 minutes walking test 2 months
  2 minutes walking test : Timing Walking test. Higher values represent a better outcome
Posturographic data (Satel Platform) variation | Change from baseline Posturographic data at 2 months
  Posturographic data test : Statokinesigram and stabilogram
Temporo-spatial parameters of gait (GAITRite walkway system) variation | Change from baseline Temporo-spatial parameters of GAITRite walkway system at 2 months
  Temporo-spatial parameters of GAITRite walkway system test : Walking test : lengh, timing and speed recorded. Higher values represent a better outcome for speed and lengh
Parkinson's Disease Questionnaire 39-item score variation | Change from baseline Parkinson's Disease Questionnaire 39-item at 2 months
  Parkinson's Disease Questionnaire 39-item test : Quality of life evaluation; 39 items quoted "never" "rarely" "sometimes" "often" or "always".
Beck Depression Inventory score variation | Change from baseline Beck Depression Inventory at 2 months
  Beck Depression Inventory test : depression evaluation . 21 items quoted 0(normal) to 3 (severe). Total score recorded : Minimum=0 Maximum = 63. Higher values represent a worse outcome
Clinical Global Impression (CGI) score variation | Change from beseline Clinical Global Impression at 2 months
  Clinical Global Impression test : Global improvement evaluation : 1 item quoted 1 (very high improvement) to 7 (very high worsening). Higher value represent a worse outcome
Isokinetic lower-limb muscle strength results variation | Change from baseline Isokinetic lower-limb muscle strength at 2 months
  Isokinetic lower-limb muscle strength test : muscular strenght evaluation. Right anf left quadriceps and harmstrings strenght evaluation. Higher values represent a better outcome
Maximal oxygen uptake (V02max) results variation | Change from baseline Maximal oxygen uptake at 2 months
  Maximal oxygen uptake test : cardio-respiratory capacity evaluation. Higher value represent a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- CH Côte Basque, Bayonne, France

IPD SHARING:
Plan to Share IPD: Yes
All IPD
Supporting Information: CSR
Time Frame: End of study :June 2023

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886